CLINICAL TRIAL: NCT05146037
Title: INTERvention With Cerebral Embolic Protection in Transcatheter Aortic Valve Implantation (INTERCEPTavi): 'Carbon-Dioxide Flushing Versus Saline Flushing of Transcatheter Aortic Valves: A Single-centre Randomised Controlled Trial'
Brief Title: INTERvention With Cerebral Embolic Protection in Transcatheter Aortic Valve Implantation (INTERCEPTavi)
Acronym: INTERCEPTavi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20HH6479
Record Dates: First submitted 2021-11-11; First posted 2021-12-06 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Stroke; Aortic Valve Stenosis; Silent Cerebral Infarct; Vascular Brain Injury
Keywords: Stroke; Aortic Valve Stenosis; Silent Cerebral Infarct; Vascular Brain Injury; TAVI; Transcatheter aortic valve implantation; Transcranial doppler; Magnetic resonance imaging; CO2; Carbon dioxide
MeSH Terms: conditions — Stroke; Aortic Valve Stenosis; Cerebrovascular Trauma

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to CO2 and Saline flushing versus saline flushing only.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and outcome assessors will be blinded to intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline flushing (Active Comparator): TAVI valves will be prepared according to instruction for use(IFU) with saline flushing only.
  Interventions: Other: Saline flushing
- CO2 and saline flushing (Experimental): TAVI valves will be flushed with CO2 and then saline as per IFU
  Interventions: Other: CO2 and saline flushing

INTERVENTIONS:
Other: CO2 and saline flushing — TAVI valves will be prepared by flushing with CO2 to displace any retained air during manufacturing and preparation. The valves will then be flushed with saline as per IFU.
  Arms: CO2 and saline flushing
Other: Saline flushing — TAVI valves will be flushed with saline only as per IFU.
  Arms: Saline flushing

SUMMARY:
The study aims to evaluate the processes of a pilot single-centre randomised controlled trial (RCT) of carbon-dioxide flushing of transcatheter aortic valves (TAVI-CO2) versus standard saline flushing of valves (TAVI-S) and assess potential neuroprotection through a number of neurological endpoints for planning of a full-sized RCT

DETAILED DESCRIPTION:
Aortic stenosis (AS) is one of the most common valve diseases and is increasing worldwide due to an ageing population. Transcatheter Aortic Valve Replacement (TAVI) is a keyhole procedure that can be done through the groin to replace the narrowed aortic valve with a new valve, avoiding the need for cardiac surgery.Improved device design and greater operator experience has improved TAVI outcomes. It has become the standard treatment option in patients who are at high risk for cardiac surgery and is now being used increasingly in lower risk patients.

Cerebrovascular accidents in TAVI patients remain a significant risk with a reported 3 - 5 % risk. Furthermore, these patients have neurovascular injury that is not clinically identifiable. Covert brain injury has been identified to occur in many surgical and cardiovascular catheter-based interventions such as TAVI and can cause vascular brain injury (VBI).

TAVI valves are manufactured in room air conditions and retain air. Studies in TEVAR (Thoracic Endovascular Aortic Repair) stent grafts have shown release of air when they are deployed in the aorta. In vitro testing of TAVI valves has shown release of air when they are deployed.

Carbon-dioxide (CO2) is 1.5 times denser than air and can displace it. It is 25 times more soluble in blood than air and does not lead to bubble formation. Hence CO2 bubble are unlikely to result in significant damage. CO2 has been used in cardiac surgery with beneficial effects. It has shown to reduce peri-procedural cerebral air embolisation and post operative cognitive dysfunction.

This study aims to look at the neuroprotective benefits of flushing TAVI valves with CO2 and saline versus saline only by reducing air embolisation.

Patients undergoing TAVI will be approached to participate in this study. After consent is obtained, patients will undergo baseline MRI, neurological and neurocognitive testing pre-TAVI. Patient will be randomised to saline only or CO2 and saline flushing of their valves. During their TAVI procedure, they will have transcranial doppler (TCD) monitoring of their middle cerebral artery (MCA) bilaterally to record cerebral embolisation. Patients will also have biomarker testing pre-TAVI, post-TAVI and 24 hours following TAVI. They will have DW-MRI brain between day 1-7 following their TAVI to look for vascular brain injury. Thus MRI will be repeated at 6-months following their TAVI. Patients will also have neurological and neurocognitive testing during their inpatient admission, at 6-weeks and 6-months outpatients.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 18 and 100 years undergoing transcatheter aortic valve implantation (TAVI) for aortic stenosis under local anaesthetic.

Exclusion Criteria:

* Patients that lack capacity to provide informed consent
* Patients that have had a stroke within 12 months
* Patients aged less than 18 years of age
* Patients that are pregnant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants suitable for recruitment for larger RCT | Duration of study, approximately 15 months
  Conduct an evaluation of the processes described in this pilot RCT for a full-scale RCT including:
  1. Screening, Recruitment and Randomisation
  2. Retention in follow-up assessments
  3. Study design for a full RCT and identification of important stratification variables
  4. Refine sample size calculation for a full RCT

SECONDARY OUTCOMES:
Incidence of Vascular Brain Injury (VBI) on Diffusion Weighted-Magnetic Resonance Imaging (DW-MRI) | Post TAVI 1-7 days and 6-months post TAVI
  Assessment of the incidence of DW-MRI detected VBI lesions following TAVI procedure. Patients will have MRI following their TAVI within 1-7 days and then at 6-months post TAVI.

OTHER OUTCOMES:
Detection of periprocedural cerebral solid and gaseous emboli | During TAVI procedure
  Document the overall rate of periprocedural cerebral solid and gaseous embolisation by transcranial doppler (TCD) monitoring during the TAVI procedure.
Neurological deficit | 6 Months
  Patients will undergo neurological assessment pre TAVI (baseline), post TAVI as inpatient, at 6-weeks and 6-months following TAVI.
Inflammatory biomarker assessing brain injury | 24 hours post TAVI
  Serial measurement of pro-inflammatory biomarkers pre-operatively, at the end of procedure and 24 hours post-operatively as a marker of brain damage including S100B
Neurocognitive decline | 6 Months
  Patients will undergo neurocognitive assessment pre TAVI (baseline), post TAVI as inpatient, at 6-weeks and 6-months following TAVI.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Mikhail, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Inci K, Koutouzi G, Chernoray V, Jeppsson A, Nilsson H, Falkenberg M. Air bubbles are released by thoracic endograft deployment: An in vitro experimental study. SAGE Open Med. 2016 Dec 7;4:2050312116682130. doi: 10.1177/2050312116682130. eCollection 2016. PMID 27994872
- [Background] Rohlffs F, Tsilimparis N, Saleptsis V, Diener H, Debus ES, Kolbel T. Air Embolism During TEVAR: Carbon Dioxide Flushing Decreases the Amount of Gas Released from Thoracic Stent-Grafts During Deployment. J Endovasc Ther. 2017 Feb;24(1):84-88. doi: 10.1177/1526602816675621. Epub 2016 Oct 26. PMID 27798380
- [Background] Martens S, Neumann K, Sodemann C, Deschka H, Wimmer-Greinecker G, Moritz A. Carbon dioxide field flooding reduces neurologic impairment after open heart surgery. Ann Thorac Surg. 2008 Feb;85(2):543-7. doi: 10.1016/j.athoracsur.2007.08.047. PMID 18222261
- [Background] Bismuth J, Garami Z, Anaya-Ayala JE, Naoum JJ, El Sayed HF, Peden EK, Lumsden AB, Davies MG. Transcranial Doppler findings during thoracic endovascular aortic repair. J Vasc Surg. 2011 Aug;54(2):364-9. doi: 10.1016/j.jvs.2010.12.063. Epub 2011 Mar 3. PMID 21371850
- [Background] Perera AH, Rudarakanchana N, Monzon L, Bicknell CD, Modarai B, Kirmi O, Athanasiou T, Hamady M, Gibbs RG. Cerebral embolization, silent cerebral infarction and neurocognitive decline after thoracic endovascular aortic repair. Br J Surg. 2018 Mar;105(4):366-378. doi: 10.1002/bjs.10718. Epub 2018 Feb 12. PMID 29431856